CLINICAL TRIAL: NCT05604456
Title: Secondary Ear Reconstructions Based on Nagata Method for Unsatisfactory Outcomes After Microtia Surgeries
Brief Title: Secondary Ear Reconstructions Based on Nagata Method
Status: Completed | Type: Observational
Sponsor: Xiaohui Su (Other)
Responsible Party: Sponsor-Investigator, Xiaohui Su, Clinical Physician, First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Other Study IDs: SERNM
Record Dates: First submitted 2022-10-28; First posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Secondary Ear Reconstructions Based on Nagata Method

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: secondary ear reconstruction based on Nagata method — Secondary auricular reconstructions based on Nagata method were conducted on patients who sought for secondary revision.

SUMMARY:
The goal of this observational study is to provide a feasible surgical strategy based on Nagata method for patients who require secondary revision surgeries and to verify its long-term aesthetic outcomes. The main question it aims to answer is:

• Whether ear reconstruction surgery based on Nagata method can improve the unsatisfactory outcomes of primary reconstruction surgery? Participants who had accepted secondary ear reconstruction based on Nagata method in our department will be required to received questionnaires in the follow-up and their photographs will be collected for reconstructed ear evaluation of its realness through convolutional neural network (CNN) models we previously developed.

ELIGIBILITY:
Inclusion Criteria:

* Chest circumference larger than 60cm at the lowest sternum level;
* Willingness to participate long-term follow-ups;
* Ability to correctly understand the questionnaire(>8 years old).

Exclusion Criteria:

* Patients with damaged superficial temporal artery (STA);
* Patients with poor condition of rib cartilage;
* Patients with active inflammation in auricular area;
* Patients who refuses surgical approach.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Microtia patients seeking for secondary ear reconstructions who had previously received reconstructive surgeries while the aesthetic outcomes were displeasing
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Preoperative and postoperative scores evaluated based on CNN | change from baseline in appearance scores at 7 months after secondary surgery
  Preoperative and postoperative photographs were acquired for reconstructed ear evaluation of its realness and appearance improvement through convolutional neural network (CNN) models we previously developed.

SECONDARY OUTCOMES:
Five-point Likert scale scores | at least 7 months after secondary surgery
  Five-point Likert scale score will be collected to show patient-reported outcomes in the follow-up study through questionnaires to assess patients' postoperative satisfaction. This questionnaire includes overall appearance, size, projection and subunits of the ear and the postoperative status of donor site. 1 = poor and 5 = excellent.

CONTACTS AND LOCATIONS:
Overall Officials: Meishui Wang, Master, Study Chair — First Affiliated Hospital of Fujian Medical University
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

REFERENCES:
- [Background] Long X, Yu N, Huang J, Wang X. Complication rate of autologous cartilage microtia reconstruction: a systematic review. Plast Reconstr Surg Glob Open. 2013 Nov 7;1(7):e57. doi: 10.1097/GOX.0b013e3182aa8784. eCollection 2013 Oct. PMID 25289252
- [Background] Akter F, Mennie JC, Stewart K, Bulstrode N. Patient reported outcome measures in microtia surgery. J Plast Reconstr Aesthet Surg. 2017 Mar;70(3):416-424. doi: 10.1016/j.bjps.2016.10.023. Epub 2016 Nov 23. PMID 28041938
- [Background] Ye J, Lei C, Wei Z, Wang Y, Zheng H, Wang M, Wang B. Evaluation of reconstructed auricles by convolutional neural networks. J Plast Reconstr Aesthet Surg. 2022 Jul;75(7):2293-2301. doi: 10.1016/j.bjps.2022.01.037. Epub 2022 Jan 31. PMID 35183463
- [Background] Reinisch JF, van Hovell Tot Westerflier CVA, Gould DJ, Tahiri YT. Secondary Salvage of the Unsatisfactory Microtia Reconstruction. Plast Reconstr Surg. 2020 May;145(5):1252-1261. doi: 10.1097/PRS.0000000000006766. PMID 32332549
- [Background] Yue X, Jiang H, Pan B, He L, Dong W, Yang Q. Secondary surgery for the unsatisfactory auricle after auricular reconstruction. Int J Pediatr Otorhinolaryngol. 2022 Mar;154:111043. doi: 10.1016/j.ijporl.2022.111043. Epub 2022 Jan 14. PMID 35063805
- [Background] Ronde EM, Esposito M, Lin Y, van Etten-Jamaludin FS, Bulstrode NW, Breugem CC. Long-term complications of microtia reconstruction: A systematic review. J Plast Reconstr Aesthet Surg. 2021 Dec;74(12):3235-3250. doi: 10.1016/j.bjps.2021.08.001. Epub 2021 Aug 17. PMID 34481742
- [Background] Varni JW, Limbers CA, Burwinkle TM. How young can children reliably and validly self-report their health-related quality of life?: an analysis of 8,591 children across age subgroups with the PedsQL 4.0 Generic Core Scales. Health Qual Life Outcomes. 2007 Jan 3;5:1. doi: 10.1186/1477-7525-5-1. PMID 17201920
- [Background] Lee TS, Lim SY, Pyon JK, Mun GH, Bang SI, Oh KS. Secondary revisions due to unfavourable results after microtia reconstruction. J Plast Reconstr Aesthet Surg. 2010 Jun;63(6):940-6. doi: 10.1016/j.bjps.2009.04.016. Epub 2009 May 17. PMID 19451041
- [Derived] Su XH, Ye J, Lei C, Wei SJ, Zheng HB, Shan XY, Wang B, Wang MS. Secondary ear reconstruction based on the Nagata method after unsatisfactory microtia surgery outcomes. J Plast Reconstr Aesthet Surg. 2023 Dec;87:251-258. doi: 10.1016/j.bjps.2023.10.075. Epub 2023 Oct 14. PMID 37924716